CLINICAL TRIAL: NCT04382976
Title: The Incidence and the Risk Factors of Nephrocalcinosis in Very Preterm Infants at the Neonatology Centre of Vilnius University Hospital Santaros Klinikos
Brief Title: The Incidence and the Risk Factors of Nephrocalcinosis in Very Preterm Infants
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Other Study IDs: 158200-R-100
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Nephrocalcinosis; Preterm Infant
MeSH Terms: conditions — Nephrocalcinosis; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess the incidence and the risk factors of nephrocalcinosis in very preterm infants using patient data collected during hospitalisation at the Neonatology Centre.

DETAILED DESCRIPTION:
Nephrocalcinosis in preterm infants develops as a result of imbalance between the factors promoting or inhibiting formation of kidney stones. It is caused by intensive treatment as well as functional and morphological kidney immaturity. There is a correlation between the prevalence of nephrocalcinosis and low gestational age.

The study aims prospectively to assess the incidence and the risk factors of nephrocalcinosis in very preterm infants less than 32 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants of the gestational age of <32 weeks;
* parental consent acquired.

Exclusion Criteria:

* death before 28 days of age;
* congenital defects;
* no kidney ultrasound results;
* no parental consent.

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population is a group of very preterm infants less than 32 weeks of gestation during hospitalisation at the Neonatology Centre.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
The incidence of nephrocalcinosis in very preterm infants less than 32 weeks of gestation | 3 years
  Kidney ultrasound results will divide preterm infants in the group with and without nephrocalcinosis (control).

SECONDARY OUTCOMES:
Compare demographic, clinical, biochemical and treatment results between nephrocalcinosis and the control (without nephrocalcinosis) groups. | 3 years
  Patients data (demographic, clinical, biochemical and treatment results) collected during hospitalisation at the Neonatology Centre will be compared between nephrocalcinosis and control group.
To evaluate the dynamics of nephrocalcinosis at 6 and 12 months of corrected age. | 6 and 12 months of corrected age
  Nephrologist consultation of the infants with nephrocalcinosis at 6 and 12 months of corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Rasa Garunkstiene, PhD, Principal Investigator — Vilnius University
Locations (1):
- Vilnius University, Neonatology Centre, Vilnius, Lithuania